CLINICAL TRIAL: NCT05133557
Title: Effects of Chewing Gum Containing Xylitol and Blackberry Extract on Oral Microbiota
Brief Title: Delivery of Polyphenols in Gum as an Anti-Caries Agent
Acronym: BBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Miller (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Craig Miller, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 12-0704-F6A; R42DE018839 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This study was a randomized, crossover-washout design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each volunteer was allocated xylitol-containing placebo gum or xylitol-containing BBE gum according to a predetermined randomization scheme. To ensure investigator blinding, test products were dispensed through other staff members who kept the assignment codes in sealed envelopes. Randomization resulted in half the participants receiving placebo gum (2 gram; 1 gram xylitol) first, and half receiving first the BBE gum (2 gram; 1 gram xylitol and 100 mg BBE) that were identical in size, shape, color and flavor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Half the participants receiving placebo gum (2 gram; 1 gram xylitol) first,
  Interventions: Other: Chewing gum containing xylitol and blackberry extract (BBE)
- BBE gum (Experimental): Half receiving first the BBE gum (2 gram; 1 gram xylitol and 100 mg BBE) that were identical in size, shape, color and flavor. After 1 week the groups cross-over and chewed the other gum.
  Interventions: Other: Chewing gum containing xylitol and blackberry extract (BBE)

INTERVENTIONS:
Other: Chewing gum containing xylitol and blackberry extract (BBE) — On the day of gum chewing, four pieces of gum were provided per the assigned group, and each volunteer was requested to chew the gum four times daily (i.e., at 9 am, 11 am, 1 pm and 3 pm). Each gum chewing interval was for 20 minutes.

SUMMARY:
The short-term effects of chewing gum containing xylitol and/or blackberry extract on oral microbiota was studied. Fifty healthy adults participated in a randomized, placebo-controlled, cross-over design study.

DETAILED DESCRIPTION:
The short-term effects of chewing gum containing xylitol and/or blackberry extract on oral microbiota was studied. Fifty healthy adults participated in a randomized, placebo-controlled, cross-over design study. One group chewed 1 piece of xylitol-containing chewing gum 4 times/day and the other chewed 1 piece of BBE+xylitol-containing gum 4 times/day. All wore a custom stent with a sterile enamel chip luted to the facial surface during the 1-day experiment. Unstimulated saliva was collected at 8 am and 4 pm, and enamel chips were harvested at 4 pm. A week later participants chewed gum from the other group. The bacterial composition in saliva and on the enamel chips were assessed using real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy, had 20 or more natural erupted teeth, and had gingivitis (bleeding on probing [BOP] in more than 15% of sites, less than 25% sites with > 4 mm probing pocket depths (PPD), and less than 5% sites with 5 mm depth PPD, who were a non-smoker, willing to participate, and verbally understood and signed an informed consent prior to enrollment

Exclusion Criteria:

* unable or unwilling to provide informed consent or follow study protocol, current smoker, systemic condition including diabetes mellitus, liver disease, kidney disease, autoimmune disease, and any cardiovascular condition that would require premedication prior to dental treatment, use of systemic antibiotics within three months of study entry, use of over the counter or prescription medications known to have anti-inflammatory/immunosuppressant activities (e.g., nonsteroidal anti-inflammatory drugs (>14 day use in past 3 months), steroids, vitamin supplements, statin drugs, topical chlorhexidine on a daily basis, pregnancy as diagnosed by administered of a pregnancy test, cancer or cancer therapy within the last year, immunosuppression (e.g., organ transplant), orthodontic therapy (current or within the last 6 months), inability to communicate verbally or in writing, clinically detectable oral mucosal inflammatory condition (e.g., aphthous, lichen planus, leukoplakia, oral cancer), or febrile illness, persistent cough or current infectious condition (e.g., influenza, hepatitis), or any PPD of 6 mm or greater at the time of the baseline periodontal examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Total salivary bacteria count | 7 hours
  Comparative difference in the total salivary bacteria count after chewing 4 pieces of gum

SECONDARY OUTCOMES:
Bacteria count on enamel | 7 hours
  Comparative difference in the total bacteria count after chewing 4 pieces of gum (placebo vs. BBE gum)

CONTACTS AND LOCATIONS:
Overall Officials: Craig S Miller, DMD, MS, Principal Investigator — University of Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavanagh HM, Hipwell M, Wilkinson JM. Antibacterial activity of berry fruits used for culinary purposes. J Med Food. 2003 Spring;6(1):57-61. doi: 10.1089/109662003765184750. PMID 12804021
- [Background] Danaher RJ, Wang C, Dai J, Mumper RJ, Miller CS. Antiviral effects of blackberry extract against herpes simplex virus type 1. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Sep;112(3):e31-5. doi: 10.1016/j.tripleo.2011.04.007. PMID 21827957
- [Background] Dai J, Patel JD, Mumper RJ. Characterization of blackberry extract and its antiproliferative and anti-inflammatory properties. J Med Food. 2007 Jun;10(2):258-65. doi: 10.1089/jmf.2006.238. PMID 17651061
- [Background] Takeuchi K, Asakawa M, Hashiba T, Takeshita T, Saeki Y, Yamashita Y. Effects of xylitol-containing chewing gum on the oral microbiota. J Oral Sci. 2018 Dec 27;60(4):588-594. doi: 10.2334/josnusd.17-0446. Epub 2018 Nov 15. PMID 30429438
- See also: UK Healthcare website — https://ukhealthcare.uky.edu/doctors/craig-miller